CLINICAL TRIAL: NCT01316016
Title: Effects of Rose Hip Intake on Risk Markers of Type 2 Diabetes and Cardiovascular Disease: a Randomized Double-blind Cross-over Investigation in Obese Persons
Brief Title: Antidiabetic Properties of Rose Hip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Cecilia Holm, Lund University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: LUAFC002
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2011-03-16 (Estimated); Status verified 2011-02

CONDITIONS: Obesity
Keywords: obesity; glucose intolerance; cholesterol; blood pressure
MeSH Terms: conditions — Obesity; Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rose hip (Experimental)
  Interventions: Dietary Supplement: Rose hip

INTERVENTIONS:
Dietary Supplement: Rose hip — 40 g of rose hip powder daily for 6 weeks.

SUMMARY:
The purpose of this study is to determine whether daily intake of a drink containing rose hip powder reduces risk markers of type diabetes and cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30
* willingness to participate in the study
* willingness to comply with the daily intake of drinks and the recommended energy intake during the course of the study

Exclusion Criteria:

* diabetes
* previous or ongoing insulin treatment
* abnormal thyroid status
* abnormal liver status
* abnormal kidney status
* known gastrointestinal disorder
* pregnancy
* suspected allergy to ingredients of the drinks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Katzman, MD/PhD, Study Chair — Lund University
Locations (1):
- Endocrinology Clinic, Lund University Hospital, Lund, Sweden

REFERENCES:
- [Background] Andersson U, Henriksson E, Strom K, Alenfall J, Goransson O, Holm C. Rose hip exerts antidiabetic effects via a mechanism involving downregulation of the hepatic lipogenic program. Am J Physiol Endocrinol Metab. 2011 Jan;300(1):E111-21. doi: 10.1152/ajpendo.00268.2010. Epub 2010 Oct 19. PMID 20959531